CLINICAL TRIAL: NCT04473053
Title: DEFINE - Evaluating Therapies for COVID-19
Acronym: DEFINE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Oxford (Other); Latus Therapeutics (Industry); Scottish National Blood Transfusion Service (SNBTS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC20063
Record Dates: First submitted 2020-07-09; First posted 2020-07-16 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — nafamostat; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomised clinical trial - currently two treatment arms and one standard of care arm. More assets will be added to the protocol as evidence emerges.
Who Masked: Outcomes Assessor
Masking Description: The biomarker analysis team will be masked to the trial treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nafamostat (Experimental): It is intended that the licensed dose (0.2mg/kg/hr) in Japan will be used. Patients randomised to Nafamostat will receive a continuous intravenous infusion at 0.2 mg/kg/hr for 7 days. If a participant is discharged from hospital or can no longer receive this treatment, the treatment will be stopped.
  Interventions: Drug: Nafamostat Mesilate
- TD139 (Experimental): Patients will inhale 5mg x 2 (10 mg) twice daily for the first 48 hrs and then subsequently 5mg x 2 (10 mg) once daily for the remaining 12 days. Unless a participant is discharged from hospital or can no longer use an inhaler - in which case treatment will be stopped at such time.
  CE marked inhalers will be provided by the Manufacturer. All patients will receive guidance on how to use the inhaler by an appropriately trained member of the research team. Two individual inhalers will be used by each patient over the course of the 14 day study period (each inhaler will be used by one patient for 7 days) and will be thoroughly cleaned with an antiseptic wipe before and after each use.
  Interventions: Drug: TD139
- Standard of Care (Active Comparator): Nafamostat and TD139 will be compared to the Standard of Care arm.
  Interventions: Other: Standard care
- Allogeneic SARS-CoV-2 VSTs (Experimental): This is an early dose escalation safety trial phase Ib/IIa interventional clinical trial with SARS-CoV-2 VSTs. This is a standalone arm of the Define study and will not be compared to any other trial appendices. A dose escalation strategy from 2x104 cells/kg to 2x106 cells/kg (based on standard 75kg weight) will be administered to patients with COVID-19 infection, and patients will be followed up to ensure their safety.
  Interventions: Biological: Allogeneic SARS-CoV-2 VSTs

INTERVENTIONS:
Drug: Nafamostat Mesilate — Nafamostat has been shown to have potential antiviral effects against MERS CoV and is thought to possibly inhibit SARS CoV2 infection via inhibition of viral entry due to inhibition of TMPRSS2. In addition, nafamostat has potent anticoagulant properties which may provide benefit in patients with DIC, a common finding in serious cases of COVID-19. Nafamostat has been broadly well tolerated in clinical trials in patients with DIC and acute pancreatitis.
  Arms: Nafamostat
Drug: TD139 — TD139 is a specific inhibitor of galectin-3 which has been investigated in healthy volunteers and patients with IPF. No serious drug related serious adverse events have been reported to date. TD139 had no impact on cardiac, haematological or biochemical measures of safety during trials in humans to date. Beneficial effects on biomarker measures of lung inflammation were observed in patients with IPF. It is the purpose of this investigation to examine the potential for delivery of this inhibitor in pre-ventilator patients hospitalised with COVID-19 to examine whether this may lead to detectable changes in blood biomarkers, reduce viral load and also reduce disease severity such as time to ventilation.
  Arms: TD139
Other: Standard care — Patients will receive standard care.
  Arms: Standard of Care
Biological: Allogeneic SARS-CoV-2 VSTs — The allogeneic SARS-CoV-2 VSTs are manufactured in a single stage process directly from the starting material procured from suitable post COVID-19 recovered individuals. This is an early dose escalation safety trial phase Ib/IIa interventional clinical trial with SARS-CoV-2 VSTs.
  Arms: Allogeneic SARS-CoV-2 VSTs

SUMMARY:
COVID-19 is a community acquired pneumonia caused by infection with a novel coronavirus, SARS CoV2 and is a serious condition with high mortality in hospitalised patients, for which there is no currently approved treatment other than supportive care. Urgent investigation of potential treatments for this condition is required.

This protocol describes an overarching and adaptive trial designed to provide safety, pharmacokinetic (PK)/ pharmacodynamic (PD) information and exploratory biological surrogates of efficacy which may support further development and deployment of candidate therapies in larger scale trials of COVID-19 positive patients receiving normal standard of care.

Given the spectrum of clinical disease, community based infected patients or hospitalised patients can be included. Products requiring parenteral administration will only be investigated in hospitalised patients. Patients will be divided into cohorts, a) community b) hospitalised patients with new changes on a chest x-ray (CXR) or a computed tomography (CT) scan or requiring supplemental oxygen and c) hospitalised requiring assisted ventilation. Participants may be recruited from all three of these cohorts, depending on the experimental therapy, its route of administration and mechanism of action. The relevant cohort(s) for any given therapy will be detailed in the therapy-specific appendix.

Candidate therapies can be added to the protocol and previous candidates removed from further investigation as evidence emerges. The trial will be monitored by an independent Data Monitoring Committee (DMC) to ensure patient safety.

Each candidate cohort will include a small cohort of patients randomised to candidate therapy or existing standard of care management dependent on disease stage at entry. Cohort numbers will be defined in the protocol appendices.

This is a Phase IIa experimental medicine trial and as such formal sample size calculations are not appropriate.

DETAILED DESCRIPTION:
This trial platform aims to support the repurposing of promising therapeutic assets with prior use in humans but without prior information on use in COVID-19, to determine the PK-PD profile of the agent, compared to standard of care supportive therapy, in small cohorts of COVID-19 patients. The results of these studies are intended to provide initial safety, pharmacokinetic and pharmacodynamic data and experimental medicine data to support further evaluation in existing national and international trial networks for candidates demonstrating appropriate impact on the dynamic marker of interest. The key interception is to mitigate the lung damage in patients with COVID-19 that leads to respiratory failure. As such, the assets in this programme will focus on abrogating putative mechanisms implicated in COVID-19 respiratory disease.

Existing approaches in clinical trials involve novel or repurposed antivirals or immunomodulatory approaches involving agents such as corticosteroids, interferon-β or hydroxychloroquine. A major limitation in the design of many early clinical trials is the limited amount of mechanistic data from patients with COVID-19. Mechanisms have been inferred from animal models, related infections or clinical syndromes. These approaches have infrequently translated to human disease. For example, remdesivir efficacy in animal models of Ebola Virus Disease (EVD) did not translate to human disease and hydroxychloroquine antiviral affects in vitro have not translated to humans against other viruses. Some drugs, such as repurposing of the anti-retroviral protease Kaletra, are still being pursued despite uncertain mechanism and despite evidence that this aspartyl protease cannot bind to the cysteine chymotrypsin-like protease that is Kaletra's putative target in COVID-19.

There is a clear and urgent need to pursue experimental medicine studies in humans to establish a solid mechanistic basis for rapid evaluation, including in existing clinical trial platforms against COVID-19 (e.g DoH RECOVERY and NIHR-CLRN industry adopted studies).

The trial will be as flexible as possible to ensure a broad range of patients can be recruited and candidate therapies can be added or removed as evidence emerges. The interim trial results will be monitored by an independent DMC to evaluate any patient safety signals.

As COVID-19 follows a variable clinical path in individual patients, the protocol is designed to enable inclusion of patients across the disease stages. The trial is intended to provide mechanistic data from patients receiving standard of care therapy and from patients treated with the therapy candidates. The study will enable delivery of pharmacokinetic information and effects of standard of care and candidate agents on surrogate biomarkers of the disease process and the specific drug target.

ELIGIBILITY:
Eligibility criteria for each arm is specified in the appendix and may vary depending on the intervention. As an example, eligibility criteria from the Nafamostat and TD139 arms has been provided:

Inclusion Criteria:

* Provision of informed consent from the patient or representative
* Aged at least 16 years
* If the patient is of child bearing potential, the patient, and their partner(s), agree to use medically-accepted double-barrier methods of contraception (eg, barrier methods, including male condom, female condom or diaphragm with spermicidal gel) during the study (if randomised to a treatment arm) and for at least 90 days after termination of study therapy. A vasectomised partner would be considered an appropriate birth control method provided that the partner is the sole male sexual partner and the absence of sperm has been confirmed.
* COVID-19 positive

Exclusion Criteria:

* Current or recent history, as determined by the Investigator, of severe, progressive, and/or uncontrolled cardiac disease (NYHA class IV), uncontrolled renal disease (eGFR <30 mL/min/1.73 m2), severe liver dysfunction (ALT/AST >5x ULN) or bone marrow failure (Hb <80 g/L AND ANC<0.5 mm3 AND platelet count <50,000 uL)
* Women who are pregnant or breastfeeding.
* Participation in another clinical trial of an investigational medicinal product (CTIMP)
* Known hypersensitivity to the IMP or excipients (e.g. lactose)
* Pre-existing or Cconcomittant use of off-label treatments for COVID-19 that are not recognised as locally approved standard care.
* Significant electrolyte disturbance (hyperkalaemia potassium >5.0 mmol/L or hyponatraemia sodium < 120mmol/L)
* Patient currently receiving potassium sparing diuretics that cannot be reasonably withheld
* Patient currently receiving prophylactic or therapeutic anticoagulantsanticoagulation or antiplatelet agents that cannot be reasonably withheld if randomised to Nafamostat
* Patients (or their partners) planning on donating sperm/eggs during the trial period
* Ongoing dialysis
* History of serious liver disease (Child Pugh score > 10)
* Hemoglobin < 80 g/L
* Any known allergy to the IMP/excipients
* Severe uncontrolled diabetes mellitus
* In the Investigator's opinion, patient is unwilling or unable to comply with drug administration plan, laboratory tests or other study procedures.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
The safety of the candidate therapies in COVID-19 patients by measuring physiological changes in the circulatory and respiratory system. | Up to 16 days post treatment
  Measure vital signs (blood pressure/heart rate/temperature and respiratory rate)
The safety of the candidate therapies in COVID-19 patients by recording the number of treatment related adverse events. | Up to 90 days post treatment
  Record number of participants With treatment-related adverse events

SECONDARY OUTCOMES:
Measuring the PK of the proposed trial treatments in COVID-19 patients. | 6 months
  Measure maximum plasma concentration [Cmax] in blood samples.
Measure a change in the expression of key coagulation biomarkers in the blood of COVID-19 patients during and after treatment period. | 6 months
  Change in expression or activity of coagulation markers in serial blood samples taken before, during and after treatment.
Measure a change in the expression of key cytokines in the blood of COVID-19 patients during and after treatment period. | 6 months
  Change in expression or activity of inflammatory cytokines in serial blood samples taken before, during and after treatment.
To evaluate the improvement or deteroriation of patients in each treatment arm. | 16 days
  Record changes in National Early Warning Score (NEWS) 2 score. Scale is from 0-20, with a higher number indicating a higher risk of morbidity.
To evaluate the number of oxygen-free days. | 16 days
  Duration (days) of oxygen use
To evaluate incidence of any form of new ventilation use. | 16 days
  Duration (days) of ventilation
To evaluate ventilator-free days | 16 days
  Duration of ventilation-free days.
  • Incidence of any form of new ventilation use and duration (days) of new ventilation use.
Change in the ratio of the oxygen saturation to fraction of inspired oxygen concentration (SpO2/FiO2) | 16 days
  SpO2/FiO2, measured daily from randomisation to Day 15, hospital discharge, or death
To evaluate SARS-CoV-2 viral load. | 15 days
  Qualitative and quantitative polymerase chain reaction (PCR) determination of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in oropharyngeal/nasal/saliva swab while hospitalised on Days 1, 3, 5, 8, 11, 15.
To evaluate time to discharge | 16 days
  Duration of total hospital stay
  • Duration to discharge following treatment
To evaluate the use of renal dialysis or haemofiltration for each treatment arm. | 16 days
  Record requirement for renal dialysis or haemofiltration

CONTACTS AND LOCATIONS:
Overall Officials: Kev Dhaliwal, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The research team actively encourage data sharing to expedite the development of COVID-19 treatments. The study team will provide data to other researchers on request and following the agreement of a data sharing plan. No confidential information regarding participants will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 90 days after data analysis has been completed for each arm. This data will be available on request and a time frame can be discussed further when required.

REFERENCES:
- [Background] Cooper RS, Fraser AR, Smith L, Burgoyne P, Imlach SN, Jarvis LM, Turner DM, Zahra S, Turner ML, Campbell JDM. Rapid GMP-Compliant Expansion of SARS-CoV-2-Specific T Cells From Convalescent Donors for Use as an Allogeneic Cell Therapy for COVID-19. Front Immunol. 2021 Jan 8;11:598402. doi: 10.3389/fimmu.2020.598402. eCollection 2020. PMID 33488592
- [Background] Gaughan E, Quinn T, Bruce A, Antonelli J, Young V, Mair J, Akram A, Hirani N, Koch O, Mackintosh C, Norrie J, Dear JW, Dhaliwal K. Evaluation of new or repurposed treatments for COVID-19: protocol for the phase Ib/IIa DEFINE trial platform. BMJ Open. 2021 Dec 15;11(12):e054442. doi: 10.1136/bmjopen-2021-054442. PMID 34911721
- [Result] Quinn TM, Gaughan EE, Bruce A, Antonelli J, O'Connor R, Li F, McNamara S, Koch O, MacKintosh C, Dockrell D, Walsh T, Blyth KG, Church C, Schwarze J, Boz C, Valanciute A, Burgess M, Emanuel P, Mills B, Rinaldi G, Hardisty G, Mills R, Findlay EG, Jabbal S, Duncan A, Plant S, Marshall ADL, Young I, Russell K, Scholefield E, Nimmo AF, Nazarov IB, Churchill GC, McCullagh JSO, Ebrahimi KH, Ferrett C, Templeton K, Rannard S, Owen A, Moore A, Finlayson K, Shankar-Hari M, Norrie J, Parker RA, Akram AR, Anthony DC, Dear JW, Hirani N, Dhaliwal K. Randomised controlled trial of intravenous nafamostat mesylate in COVID pneumonitis: Phase 1b/2a experimental study to investigate safety, Pharmacokinetics and Pharmacodynamics. EBioMedicine. 2022 Feb;76:103856. doi: 10.1016/j.ebiom.2022.103856. Epub 2022 Feb 11. PMID 35152152
- [Result] Gaughan EE, Quinn TM, Mills A, Bruce AM, Antonelli J, MacKinnon AC, Aslanis V, Li F, O'Connor R, Boz C, Mills R, Emanuel P, Burgess M, Rinaldi G, Valanciute A, Mills B, Scholefield E, Hardisty G, Findlay EG, Parker RA, Norrie J, Dear JW, Akram AR, Koch O, Templeton K, Dockrell DH, Walsh TS, Partridge S, Humphries D, Wang-Jairaj J, Slack RJ, Schambye H, Phung D, Gravelle L, Lindmark B, Shankar-Hari M, Hirani N, Sethi T, Dhaliwal K. An Inhaled Galectin-3 Inhibitor in COVID-19 Pneumonitis: A Phase Ib/IIa Randomized Controlled Clinical Trial (DEFINE). Am J Respir Crit Care Med. 2023 Jan 15;207(2):138-149. doi: 10.1164/rccm.202203-0477OC. PMID 35972987
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343